CLINICAL TRIAL: NCT00025818
Title: Six Month Clinical Research Study for Patients With Moderate or Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192371-011-01
Record Dates: First submitted 2001-10-26; First posted 2001-10-29 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Keratoconjunctivitis Sicca; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Scleroderma, Systemic
Keywords: dry eyes; rheumatoid arthritis; Lupus; Sjogren's syndrome; myositis; scleroderma; autoimmune disorder
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Scleroderma, Systemic; Dry Eye Syndromes; Myositis; Scleroderma, Diffuse; Autoimmune Diseases

INTERVENTIONS:
Drug: Ophthalmic Emulsion

SUMMARY:
A six-month clinical research trial to evaluate the effectiveness of an investigational medication for the treatment of dry eye syndrome in patients that have been diagnosed with moderate to severe dry eye syndrome, an autoimmune disorder AND/OR females 65 years of age or older.

ELIGIBILITY:
* Eighteen years or older
* Diagnosis of moderate to severe dry eyes for at least 6 months and meet one or all of the following criteria:
* Diagnosis of autoimmune disorder
* Female 65 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2001-05; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Eyecare of La Jolla, La Jolla, California
  - UCLA, Los Angeles, California
  - Opticare, Waterbury, Connecticut
  - Brandon Eye Clinic, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - UIC Eye Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Hunkleler Eye Center, Overland Park, Kansas
  - D'Ambrosio Eye Care, Leominster, Massachusetts
  - Great Lakes Eye Institute, Saginaw, Michigan
  - Cornea Consultants of Albany, Albany, New York
  - Dr. Freedman's Office, Brooklyn, New York
  - Dr. Wittpen's Office, Stony Brook, New York
  - The Cole Eye Institute, Cleveland, Ohio
  - Northwest Cornea, Portland, Oregon
  - Corona Research, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas